CLINICAL TRIAL: NCT04342182
Title: Convalescent Plasma Therapy From Recovered Covid-19 Patients as Therapy for Hospitalized Patients With Covid-19
Brief Title: Convalescent Plasma as Therapy for Covid-19 Severe SARS-CoV-2 Disease (CONCOVID Study)
Acronym: ConCoVid-19
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: new insights into COVID19 pathogenesis
Sponsor: Erasmus Medical Center (Other)
Collaborators: Prothya Biosolutions (Industry)
Responsible Party: Principal Investigator, Bart Rijnders, MD, PhD, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL73489.078.20
Record Dates: First submitted 2020-03-31; First posted 2020-04-10 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This trial is a randomized comparative trial. Patients will be randomized between the infusion of 300mL of convP versus the standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Convalescent plasma (Experimental): Standard of care plus 300mL of convalescent plasma from COVID-19 recovered donors
  Interventions: Biological: Convalescent plasma
- Standard of care (No Intervention): standard of care (supportive care, oxygen, antibiotics)

INTERVENTIONS:
Biological: Convalescent plasma — Infusion of plasma retrieved from donors with a history of PCR proven symptomatic COVID.
  Plasma will be administered according to the Erasmus MC KIS protocol regarding the use of blood products
  Arms: Convalescent plasma

SUMMARY:
Passive immunization with immunoglobulins is occasionally used as therapy for the treatment of viral infectious diseases. Immunoglobulins are used for the treatment of CMV disease, and is effective as prophylaxis when given soon after exposure to varicella zoster virus, rabies, and hepatitis B virus.

Neutralizing antibodies against MERS, SARS-CoV-1 and SARS-CoV-2 have been shown to be present in patients previously infected with MERS, SARS-CoV-1 and SARS-CoV-2 respectively. During the 2003 SARS outbreak in Hong-Kong,a non-randomized study in hospitalized SARS patients showed that treatment with convalescent plasma (convP) from SARS-recovered donors significantly increased the day 22 discharge rate and decreased mortality. A study in non-human primates showed that rhesus macaques could not be re-infected with SARS-CoV-2 after primary infection.

With no proven effective therapy against COVID, this study will evaluate the safety and efficacy of convalescent plasma from COVID-recovered donors as a treatment for hospitalized patients with symptomatic COVID-19. The study will focus on patients who tested positive for SARS-CoV-2 in the last 96 hours before inclusion

Primary objectives

• Decrease overall mortality in patients within COVID disease

Study design:

This trial is a randomized comparative trial. Patients will be randomized between the infusion of 300mL of convP with standard of care.

Patient population:

Patients with PCR confirmed COVID disease, age >18 years Donors will be included with a known history of COVID who have been asymptomatic for at least 14 days.

Intervention: 300mL of convP Duration of treatment: ConvP will be given as a one-time infusion Duration of follow up: For the primary endpoint: until discharge or death before day 60, whichever comes first. For the secondary endpoints (with separate consent) up to 1 year.

Target number of patients: 426 Target number of donors: 100 Expected duration of accrural: 36 months

DETAILED DESCRIPTION:
Secondary (exploratory) objectives

* Evaluate the effect of 300ml convP on hospital stay
* Evaluate the change of the 8-point WHO COVID19 disease severity scale on day 15 and 30
* Evaluate the change of the 8-point WHO COVID19 disease severity scale on day 15 in the subgroup of patients with a baseline neutralizing antibody titer (PRNT50) <80
* Evaluate the effect of 300ml convP on mortality in patients admitted to the ICU
* Evaluate the effect of 300ml plasma therapy on hospital days for patients admitted to the ICU within 24 hours after admission
* Evaluate the impact of plasma therapy on the decrease in SARS-CoV2 shedding from airways
* Evaluate the difference in effect of convP on mortality in patients with a duration of symptoms < or > the median duration of symptoms in the study population
* Evaluate the impact of CTL and NK cell immunity on the likelihood of being protected from immune serum transfer
* Safety of convP therapy
* Evaluate the impact of covP on long-term lung function

ELIGIBILITY:
Inclusion Criteria:

* Patients with PCR confirmed COVID disease
* Admitted to the hospital
* The most recent PCR positive sample is <96hrs old
* Written informed consent by patient or legal patient representative
* Age at least 18 years

Exclusion Criteria:

* Participation in another intervention trial on the treatment of COVID-19 that falls under the Dutch law human research (WMO) and in which individual patients are randomized to different treatment options
* Known IgA deficiency
* Invasive ventilation for already >96 hours

Donors: Eligibility for plasma donation

Inclusions Criteria:

* A history of COVID infection that was documented by PCR
* Known ABO-Resus(D) blood group
* A screening for irregular antibodies with a titer ≤ 1:32
* Asymptomatic for at least 14 days
* Written informed consent regarding the plasmapheresis procedure
* Tested negative for HIV, HBV, HCV, HEV, HTLV and syfilis

Exclusion Criteria:

* Age <18 years and > 65 years
* Weight <50kg
* Medical history of heart failure
* History of transfusion with red blood cells, platelets or plasma
* History of organ- or tissue transplant
* A cumulative stay in the United Kingdom of ≥ 6 months in the period between 01-01-1980 and 31-12-1996
* A history of i.v. drug use
* Insulin dependent diabetes
* An underlying severe chronic illness (i.e. history of heart failure, cancer or stroke)
* Tested positive for HLA- or HNA-antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Overall mortality until discharge from the hospital or a maximum of 60 days after admission whichever comes first | until hospital discharge or a maximum of 60 days whichever comes first
  the mortality in the 300ml convP group will be compared with the control arm

SECONDARY OUTCOMES:
Impact of 300ml convP therapy on hospital days | until hospital discharge or a maximum of 60 days whichever comes first
  the hospital days in the 300ml convP group will be compared with the control arm
Impact of 300ml convP on weaning from oxygen therapy | until hospital discharge or a maximum of 60 days whichever comes first
  A patient will be considered weaned from oxygen therapy when the patient did not receive oxygen for at least 24 hours.
Impact of 300ml convP on overall mortality in patients admitted to the ICU within 24 hours after admission | until hospital discharge or a maximum of 60 days whichever comes first
  the overall mortality in hospital days in patients admitted tot the ICU within 24 hours after admission in the 300ml convP group will be compared with the patients admitted tot the ICU within 24 hours after admission in the control arm
Difference in the effect of convP on mortality in patients with a duration of symptoms less or more the median duration of symptoms in the study population | hospital discharge or a maximum of 60 days whichever comes first
  The mortality in patients with a duration of symptoms less than the median duration of symptoms in the study population will be compared with the mortality in patients with a duration of symptoms more than the median duration of symptoms in the study population
Impact of 300ml convP therapy on ICU days in patients admitted to the ICU within 24 hours after admission | Until hospital discharge, estimated average 4 weeks
  the ICU days in hospital days in patients admitted to the ICU within 24 hours after admission in the 300ml convP group will be compared with the patients admitted tot the ICU within 24 hours after admission in the control arm
Impact of plasma therapy on the decrease in SARS-CoV2 shedding from airways | until hospital discharge, estimated average 2 weeks
  airway samples will be taken on day 1 - 3 - 5 - 7 - 10 - 14 - and at discharge
Impact of CTL and NK cell immunity on the likelihood of being protected from immune serum transfer | until hospital discharge, extimated average 2 weeks
  Blood wil be drawn at day 1, day 7 and day 14
Safety of convP therapy | until hospital discharge or a maximum of 60 days whichever comes first
  Evaluation of Severe Adverse Events and transfusion related adverse events
Change of the 8-point WHO COVID19 disease severity scale on day 15 | until day 15
  The WHO COVID19 disease severity scale on day 15 will be compared with the WHO COVID19 disease severity scale on day 1
Change of the 8-point WHO COVID19 disease severity scale on day 30 | until day 30
  The WHO COVID19 disease severity scale on day 30 will be compared with the WHO COVID19 disease severity scale on day 1 and day 15
Change of the 8-point WHO COVID19 disease severity scale on day 15 in the subgroup of patients with a baseline neutralizing antibody titer (PRNT50) <80. | until day 15
  The WHO COVID19 disease severity scale on day 15 will be compared with the WHO COVID19 disease severity scale on day 1 in patients with a baseline neutralizing antibody titer (PRNT50) <80.
Impact of plasma therapy on risk of long-term structural lung damage and lung function | up to 12 months after plasma transfusion
  Low dose CT and lung function is done 6 weeks after discharge and if abnormal again 3 months after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Bart Rijnders, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (18):
- Netherlands (18):
  - Erasmus Medical Center, Rotterdam, South Holland
  - NoordWest Ziekenhuisgroep, Alkmaar
  - Onze Lieve Vrouwen Gasthuis, Amsterdam
  - Rijnstate Ziekenhuis, Arnhem
  - Reinier de Graaf Gasthuis, Delft
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Groene Hart Ziekenhuis, Gouda
  - Martini Hospital, Groningen
  - Spaarna Gasthuis, Haarlem
  - Alrijne Ziekenhuis, Leiderdorp
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Canisius-Wilhelmina Hospital, Nijmegen
  - Maasstad Ziekenhuis, Rotterdam
  - ZorgSaam Hospital, Terneuzen
  - Haaglanden Medisch Centrum, The Hague
  - Bernhoven Hospital, Uden
  - VieCuri, Venlo

REFERENCES:
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub6. PMID 37162745
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 Feb 1;2(2):CD013600. doi: 10.1002/14651858.CD013600.pub5. PMID 36734509
- [Derived] Piechotta V, Iannizzi C, Chai KL, Valk SJ, Kimber C, Dorando E, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 20;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub4. PMID 34013969
- [Derived] Chai KL, Valk SJ, Piechotta V, Kimber C, Monsef I, Doree C, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2020 Oct 12;10:CD013600. doi: 10.1002/14651858.CD013600.pub3. PMID 33044747